CLINICAL TRIAL: NCT05480033
Title: The Effect of Imagery Technique on Self-Effectiveness-Efficacy and Anxiety Levels of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Collaborators: GÜLAY YILMAZ (Unknown); BETÜL KUŞ (Unknown)
Responsible Party: Principal Investigator, Ozlem Sahin Akboga, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Imagery
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Self Efficacy; Nurse's Role
Keywords: Anxiety; Self Efficacy; Nursing students
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Imagination is linked to human creativity. Imagery is how we animate and design an object, situation and/or entity by redefining it and concretising it in our minds. In other words, imagery is the ability to create an idea or image in our minds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The imagery technique was applied to the students in this group on the day of the laboratory practice, before the lesson, once a week for 4 weeks. The laboratory practice consisted of 6 weeks. Pre-test was performed on the first week, followed by 4 weeks of imagery technique, and the pre-test was performed on the final week. In each application of the imagery technique, four scenarios that could be encountered in clinical practice that required skill practice were used for 30 minutes. The imagery technique was applied by the second author who had expertise and training in nursing and imagery technique. The stages of the imagery technique included preparation of a suitable environment, preparation of the students, setting the background music (ney sound), relaxation, focusing on the technique, visualising the situation to be imagined, loading positive and constructive expressions on the individual, distracting the student from the imagined situation, relaxation and ending the session.
  Interventions: Behavioral: Imagery Technique
- Control group (No Intervention): No intervention was performed on the students in this group.

INTERVENTIONS:
Behavioral: Imagery Technique — The stages of the imagery technique included preparation of a suitable environment, preparation of the students, setting the background music (ney sound), relaxation, focusing on the technique, visualising the situation to be imagined, loading positive and constructive expressions on the individual, distracting the student from the imagined situation, relaxation and ending the session.
  Arms: Intervention group

SUMMARY:
To determine the effect of the imagery technique used in the Nursing Fundamentals course on the self-effectiveness-efficacy and anxiety levels of students. This study was designed as a randomized controlled trial. The research was completed with a total of 85 students, 40 of which were in the intervention group and 45 in the control group. The imagery technique was applied to the intervention group once a week for 4 weeks before the laboratory practice lesson. This study are self-efficacy-sufficiecy and state and trait anxiety levels obtained from the questionnaire before and after the application. While there was no difference in the mean scores of self-efficacy-sufficiecy and trait anxiety of the students before and after the application of the imagery technique (p=0.515, p=0.456), it was determined that the mean score of state anxiety of the students in the intervention group decreased significantly after the application (p=0.044). Academic nurses should work on increasing self-efficacy and reducing the level of trait anxiety, in addition to the supportive imagery technique during training.

DETAILED DESCRIPTION:
Nursing students need to be prepared and supported to tackle problems that they are likely to experience in the future. With this in mind, this research was conducted to determine the effect of imagery technique applied in practical courses on the self-effectiveness-efficacy and anxiety levels of the nursing students.

This research was designed as a randomised controlled experimental study. The research included intervention (40 students) and control (45 students) groups, and a pre-test and post-test was applied.

The research was conducted between February 2021 and May 2021 with second-year students in the Nursing Department of the Faculty of Health Sciences of a state university in Turkey.

Interventions: The students were informed about the purpose and scope of the study and the intervention. Students who volunteered to participate in the study were randomised into groups. Afterwards, 'Personal Information Form', 'Self-Effectiveness-Efficacy Scale' and 'State-Trait Anxiety Inventory' were distributed to all students as the pre-test.

Intervention group: The imagery technique was applied to the students in this group on the day of the laboratory practice, before the lesson, once a week for 4 weeks. The laboratory practice consisted of 6 weeks. Pre-test was performed on the first week, followed by 4 weeks of imagery technique, and the pre-test was performed on the final week. In each application of the imagery technique, four scenarios that could be encountered in clinical practice that required skill practice were used for 30 minutes (Table 1).

The imagery technique was applied by the second author who had expertise and training in nursing and imagery technique. The stages of the imagery technique included preparation of a suitable environment, preparation of the students, setting the background music (ney sound), relaxation, focusing on the technique, visualising the situation to be imagined, loading positive and constructive expressions on the individual, distracting the student from the imagined situation, relaxation and ending the session.

Control group: No intervention was performed on the students in this group. After the post-test, students in the control group were shown a video on imagery technique so that they would not feel excluded and less competent and also to reduce the possible bias among the students.

This study are self-efficacy-sufficiecy and state and trait anxiety levels obtained from the questionnaire before and after the application. While there was no difference in the mean scores of self-efficacy-sufficiecy and trait anxiety of the students before and after the application of the imagery technique (p=0.515, p=0.456), it was determined that the mean score of state anxiety of the students in the intervention group decreased significantly after the application (p=0.044).

The results of this study show that the imagery technique resulted in a significant decrease in the state anxiety levels of the nursing students, while the trait anxiety and self-effectiveness-efficacy levels were not affected. There are only limited studies in the literature evaluating the effectiveness of imagery technique in basic skill practice training of the nursing students. Therefore, the results of this study are expected to contribute to the nursing profession.

ELIGIBILITY:
Inclusion Criteria:

* Students who volunteered to participate in the study,

Exclusion Criteria:

* Who do not participate in the entire application, Students who did not focus on the study were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Self-Effectiveness-Efficacy Scale | 3 MONTHS
  self-confidence
State-Trait Anxiety Inventory | 3 MONTHS
  stress levels

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No